CLINICAL TRIAL: NCT07303452
Title: A Multi-center Proof-of-concept Study to Assess the Safety and Effectiveness of the Restera™ Serene™ System When Stimulating the Hypoglossal Nerve Alone or the Hypoglossal Nerve Plus the Ansa Cervicalis Nerve for the Treatment of Obstructive Sleep Apnoea in Adult Participants.
Brief Title: Evaluation of the Restera™ Serene™ System in Adults With Obstructive Sleep Apnea
Acronym: REST-HGN+AC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Restera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM-010
Record Dates: First submitted 2025-11-28; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Target (Experimental)
  Interventions: Device: Neurostimulation
- Dual Target (Experimental)
  Interventions: Device: Neurostimulation

INTERVENTIONS:
Device: Neurostimulation — Neurostimulation via Restera Serene System

SUMMARY:
The purpose of this multi-center proof-of-concept safety and efficacy study is to collect chronic sleep-related data following percutaneous placement of electrode arrays near the hypoglossal nerve and the ansa cervicalis in adults with obstructive sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) ≤ 32 kg/m2
* AHI between 15-65 events/hour
* Participants who have either not tolerated, have failed or refused positive airway pressure (PAP)

Exclusion Criteria:

* Pregnancy or breast-feeding
* Significant upper airway anatomic abnormalities
* Significant positionally-dependent OSA
* Participants taking medications that may alter body weight

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Safety of the Restera Serene System | 6 months
  Incidence of device and/or procedure-related serious adverse events
Effectiveness of the Restera Serene System | 6 months
  Change from baseline in the Apnea-Hypopnea Index

SECONDARY OUTCOMES:
Long-term Safety of the Restera Serene System | 36 months
  Incidence of device and/or procedure-related serious adverse events
Long-term Effectiveness of the Restera Serene System | 36 months
  Change from baseline in the Apnea-Hypopnea Index

CONTACTS AND LOCATIONS:
Locations (1):
- University of Western Australia, Perth, Australia

IPD SHARING:
Plan to Share IPD: Undecided